CLINICAL TRIAL: NCT03860259
Title: The Effect of Auriculotherapy for Post-Operative Pain Management Following Rotator Cuff Surgery: A Randomized, Placebo-Controlled Study
Brief Title: Auriculotherapy for Surgical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor of Anesthesiology (with Tenure) and Orthopedic Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO18050099
Record Dates: First submitted 2019-01-22; First posted 2019-03-01 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Acute Pain; Surgery; Shoulder Pain
Keywords: opioids; auriculotherapy; acute pain; shoulder surgery
MeSH Terms: conditions — Acute Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The only person unblinded to treatment allocation will be the Principal investigator or designee -- the individual performing cryopuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Auriculotherapy without nitrogen gas (Placebo Comparator): Auriculotherapy will be performed by certified research staff using a cryopuncture device in the post-anesthesia recovery room with an empty cryopuncture with no nitrogen gas. The patient will receive an interscalene nerve block, standard of care treatment for surgery, post-operative pain management, and physical therapy.
  Interventions: Device: Auriculotherapy cryopuncture device without nitrogen gas
- Auriculotherapy with nitrogen gas (Active Comparator): Auriculotherapy will be performed by certified research staff using a cryopuncture device in the post-anesthesia recovery room with nitrogen gas. The patient will receive an interscalene nerve block, standard of care treatment for surgery, post-operative pain management, and physical therapy.
  Interventions: Device: Auriculotherapy cryopuncture device with nitrogen gas

INTERVENTIONS:
Device: Auriculotherapy cryopuncture device without nitrogen gas — Auriculotherapy cryopuncture device without nitrogen gas will be administered. In addition, an interscalene block will be performed as well as standard of care treatment for surgery, post-operative pain management and physical therapy
  Arms: Auriculotherapy without nitrogen gas
Device: Auriculotherapy cryopuncture device with nitrogen gas — Auriculotherapy cryopuncture device with nitrogen gas will be administered. In addition, an interscalene block will be performed as well as standard of care treatment for surgery, post-operative pain management and physical therapy
  Arms: Auriculotherapy with nitrogen gas

SUMMARY:
The current opioid epidemic has led to a renewed interest in exploring non-pharmacological techniques to treat post-operative pain. An increasing number of patients are suffering from the adverse effects of opioid use following surgery, including post-operative nausea and vomiting, respiratory depression, immunosuppression, constipation, and most recently, addiction. In the United States, over $600 billion is spent every year on opioid addiction, including $79 billion related to opioid addiction following surgery. Despite many initiatives to decrease the use of opiates in the preoperative setting, opioids continue to be regularly prescribed before, during and after surgery. Although the risk of opioid addiction following surgery is recognized, the percentage of patients becoming addicted to opioids following surgery is not well understood.

To date, there has been virtually no agreement regarding the duration and dosage that qualify for opioid dependence following surgery, nor that a clear estimation of the factors such as biological, psychosocial and socioeconomic that increase the risk of using opioids for extended periods of time after surgery. The interscalene block is the gold standard for postoperative pain management following shoulder surgery. However, the duration of the block does not cover rehabilitation, and in most cases, patients are discharged from the hospital with an opioid prescription. Therefore, there is a growing need to investigate complementary pain-management methods that offer a non-pharmacological solution to managing post-operative pain. Auriculotherapy is such a technique that has been shown in previous studies to provide significant analgesia without the adverse effects of opioids or other pain-relieving medications. Auriculotherapy has been shown to reduce the need for opioid immediately after surgery. However, everyone agrees that more research is needed, especially due to the concern of the placebo effect when using a needle and electro-stimulation. This study is purposely based on the use of a cryopuntor device, which has been shown to produce the same effect as needles. This is a novel complementary approach to reducing the persistence of opioid prescription following rotator cuff surgery, which is considered a model of severe functional pain. Data obtained from this study will support a future NIDA proposal to expand the use of auriculotherapy for perioperative management of pain and functional recovery associated with surgery. The use of an auriculotherapy approach has the potential of providing effective non-opioid analgesia to patients not only undergoing rotator cuff surgery, but also other surgical models.

DETAILED DESCRIPTION:
Once patient has signed the Informed Consent to participate in this trial, demographic information and medical history will be collected from each participant on the day of surgery. Research staff will record this information from the medical chart. The Medical Outcomes Study Questionnaire 12-Item Short Form Health Survey (SF-12) will also be administered at this time to obtain baseline value. Randomization will occur by assigning the participant a subject ID number, and this ID number will correspond to a treatment allocation based on a pre-designed randomization schema. This treatment allocation (intervention/control) will be contained in a sealed, opaque, envelope with the subject ID number that is designated on envelope. The master randomization list will be created and held by an independent data monitor who will both create and hold the master randomization list.

Study coordinators, Co-Is and subjects will be blinded. Only the research staff completing the treatment will be unblinded. Once the patient is randomized to a treatment group by research staff, Auriculotherapy will be performed by certified research staff using a cryoauriculopuncture in the post-anesthesia recovery room, either with nitrogen gas (intervention group), or an empty cryoauriculopunture with no gas (control group).

After proper disinfection of the designated ear, the treatment consists of the stimulation of 9 ear points on the ipsilateral ear. These points include:-Ω2 (the master point for the mesoderm), the shoulder point, 6 points involved with the pain pathway (the stellar ganglion, the sensory and motor C7 branches, the sensory master point (MSP), the reticular master point (RMP) and the point corresponding to the Thalamus). Finally, the stimulation of the ACTH point completes the treatment. The total time required to complete auriulotherapy treatment is approximately 10 minutes. The enrolled subject will also receive a pre-operative interscalene block as per standard of care. The patient will receive standard of care treatment for surgery, post-operative pain management, and physical therapy. After surgery, the subject will be assessed at time of hospital discharge to review how to complete the subject diary, administer pain satisfaction questionnaire (0-6) and obtain NRS pain at rest and with movement scores (0-10). When the patient is discharged from the hospital, the subject will be asked to take home and complete a subject diary where they will record their total narcotic/pain medication consumption, pain satisfaction score (0-6), and NRS pain score (0-10), and adverse events daily for first 5 days post-discharge. The subject will be instructed to complete the diary just before bedtime on these post-op days. The patient will be contacted via telephone on Day 5 post-operatively as a reminder to return pain diary. On post-operative Day 14, 30, 60 and 90 telephone calls, functional recovery will be measured using the Medical Outcomes Study Questionnaire 12-Item Short Form Health Survey (SF-12). The subject will also be asked to assess their overall patient satisfaction at the Day 90 call, on a scale of 0 (least satisfaction) to 10 (most satisfaction). Analgesic efficacy in both groups will also be evaluated by the amount of total narcotic consumption (measured with oral morphine equivalent doses of analgesics used to provide pain relief). Secondary outcome measures will include pain at rest and with movement, total non-narcotic pain medication consumption for the first 5-days post-discharge, time to readiness for discharge from PACU, time to hospital discharge, readmission to the hospital because of pain related issues, incidence of postoperative complications, overall patient satisfaction, patient satisfaction relating to pain management and functional recovery. Functional recovery will be measured using the Medical Outcomes Study Questionnaire 12-Item Short Form Health Survey (SF-12).

Since, starting the study, the secondary outcome measure of "Change in post-operative opioid consumption in opioid naïve subjects undergoing rotator cuff surgery" has been removed as this is repetitive of the data collected as part of the primary outcome measure and its analysis. Additionally the outcome of "Pain scores following rotator cuff surgery" was further specified to Post-operative pain at rest and Post-operative pain with movement for clarification and analysis of each individually. This was also altered from a primary to secondary outcome to match the current IRB approved protocol for this study in which pain scores were a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than 18 years of age
2. Subject is willing and able to provide informed consent
3. Subject is scheduled to undergo elective rotator cuff surgery
4. Subject has consented to an interscalene block

Exclusion Criteria:

1. Opioid dependence
2. Any subject diagnosed with a chronic pain condition which daily opioid use is needed
3. Anatomical malformation, which in the investigator's opinion may interfere with the placement of the nerve block
4. Raynaud's disease diagnosis
5. Vasculopathy
6. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alimi D., Geissmann A., Gardeur D., Bahr F. Study in fMRI of the stimulation of the auricular areas of the knee as the French -German and Chinese localizations. The Journal of Radiology. Photon 2014; 125, 133-14.
- [Background] Alimi D, Rubino C, Pichard-Leandri E, Fermand-Brule S, Dubreuil-Lemaire ML, Hill C. Analgesic effect of auricular acupuncture for cancer pain: a randomized, blinded, controlled trial. J Clin Oncol. 2003 Nov 15;21(22):4120-6. doi: 10.1200/JCO.2003.09.011. PMID 14615440
- [Background] Cho ZH, Oleson TD, Alimi D, Niemtzow RC. Acupuncture: the search for biologic evidence with functional magnetic resonance imaging and positron emission tomography techniques. J Altern Complement Med. 2002 Aug;8(4):399-401. doi: 10.1089/107555302760253577. No abstract available. PMID 12230898
- [Background] Usichenko TI, Dinse M, Hermsen M, Witstruck T, Pavlovic D, Lehmann C. Auricular acupuncture for pain relief after total hip arthroplasty - a randomized controlled study. Pain. 2005 Apr;114(3):320-327. doi: 10.1016/j.pain.2004.08.021. PMID 15777857
- [Background] Usichenko TI, Kuchling S, Witstruck T, Pavlovic D, Zach M, Hofer A, Merk H, Lehmann C, Wendt M. Auricular acupuncture for pain relief after ambulatory knee surgery: a randomized trial. CMAJ. 2007 Jan 16;176(2):179-83. doi: 10.1503/cmaj.060875. PMID 17224599
- [Background] Wetzel B, Pavlovic D, Kuse R, Gibb A, Merk H, Lehmann C, Wendt M, Usichenko TI. The effect of auricular acupuncture on fentanyl requirement during hip arthroplasty: a randomized controlled trial. Clin J Pain. 2011 Mar-Apr;27(3):262-7. doi: 10.1097/AJP.0b013e3181fd516c. PMID 21346689
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Kukreja P, Avila A, Northern T, Dangle J, Kolli S, Kalagara H. A Retrospective Case Series of Pericapsular Nerve Group (PENG) Block for Primary Versus Revision Total Hip Arthroplasty Analgesia. Cureus. 2020 May 19;12(5):e8200. doi: 10.7759/cureus.8200. PMID 32572357
- [Background] Crockett SD, Greer KB, Heidelbaugh JJ, Falck-Ytter Y, Hanson BJ, Sultan S; American Gastroenterological Association Institute Clinical Guidelines Committee. American Gastroenterological Association Institute Guideline on the Medical Management of Opioid-Induced Constipation. Gastroenterology. 2019 Jan;156(1):218-226. doi: 10.1053/j.gastro.2018.07.016. Epub 2018 Oct 16. No abstract available. PMID 30340754
- [Background] Farmer AD, Drewes AM, Chiarioni G, De Giorgio R, O'Brien T, Morlion B, Tack J. Pathophysiology and management of opioid-induced constipation: European expert consensus statement. United European Gastroenterol J. 2019 Feb;7(1):7-20. doi: 10.1177/2050640618818305. Epub 2018 Dec 14. PMID 30788113
- [Background] Kozub E, Uttermark A, Skoog R, Dickey W. Preventing Postoperative Opioid-Induced Respiratory Depression Through Implementation of an Enhanced Monitoring Program. J Healthc Qual. 2022 Jan-Feb 01;44(1):e7-e14. doi: 10.1097/JHQ.0000000000000322. PMID 34469926
- [Background] Warrender WJ, Syed UAM, Hammoud S, Emper W, Ciccotti MG, Abboud JA, Freedman KB. Pain Management After Outpatient Shoulder Arthroscopy: A Systematic Review of Randomized Controlled Trials. Am J Sports Med. 2017 Jun;45(7):1676-1686. doi: 10.1177/0363546516667906. Epub 2016 Oct 13. PMID 27729319
- [Background] Karst M, Winterhalter M, Munte S, Francki B, Hondronikos A, Eckardt A, Hoy L, Buhck H, Bernateck M, Fink M. Auricular acupuncture for dental anxiety: a randomized controlled trial. Anesth Analg. 2007 Feb;104(2):295-300. doi: 10.1213/01.ane.0000242531.12722.fd. PMID 17242083
- [Background] Lux EA, Wahl G, Erlenwein J, Wiese C, Wirz S. [Is supplemental ear acupuncture for surgical tooth removal with local anesthesia effective? : A pilot study]. Schmerz. 2017 Oct;31(5):489-498. doi: 10.1007/s00482-017-0212-3. German. PMID 28315017
- [Background] Li WS, Wan LS, Liu XJ, Li WY, Xiao JB, Zhao WX. [Effect of assisted anesthesia of auricular point magnetic sticking on postoperative recovery of gynecological surgery]. Zhongguo Zhen Jiu. 2013 Jul;33(7):648-52. Chinese. PMID 24032205
- [Background] Zhang LH, Cao CL, Li JZ, Chen ML, Wang MS, Dai CY. [Influence of auricular point sticking on incidence of nausea and vomiting and analgesia effect after gynecological laparoscopy]. Zhongguo Zhen Jiu. 2013 Apr;33(4):339-41. Chinese. PMID 23819241
- [Background] Zhang WF, Sun M, Da LM. [Electroacupuncture at auricular points for 43 cases of postpartum depression]. Zhongguo Zhen Jiu. 2012 Dec;32(12):1075-6. No abstract available. Chinese. PMID 23301469
- [Background] Usichenko T, Hacker H, Lotze M. Transcutaneous auricular vagal nerve stimulation (taVNS) might be a mechanism behind the analgesic effects of auricular acupuncture. Brain Stimul. 2017 Nov-Dec;10(6):1042-1044. doi: 10.1016/j.brs.2017.07.013. Epub 2017 Aug 2. PMID 28803834
- [Background] Vieira A, Reis AM, Matos LC, Machado J, Moreira A. Does auriculotherapy have therapeutic effectiveness? An overview of systematic reviews. Complement Ther Clin Pract. 2018 Nov;33:61-70. doi: 10.1016/j.ctcp.2018.08.005. Epub 2018 Aug 23. PMID 30396628
- [Background] Baker TE, Chang G. The use of auricular acupuncture in opioid use disorder: A systematic literature review. Am J Addict. 2016 Dec;25(8):592-602. doi: 10.1111/ajad.12453. Epub 2016 Nov 2. PMID 28051842
- [Background] Asher GN, Jonas DE, Coeytaux RR, Reilly AC, Loh YL, Motsinger-Reif AA, Winham SJ. Auriculotherapy for pain management: a systematic review and meta-analysis of randomized controlled trials. J Altern Complement Med. 2010 Oct;16(10):1097-108. doi: 10.1089/acm.2009.0451. PMID 20954963
- [Background] Contim CLV, Santo FHDE, Moretto IG. Applicability of auriculotherapy in cancer patients: an integrative literature review. Rev Esc Enferm USP. 2020 Sep 7;54:e03609. doi: 10.1590/S1980-220X2019001503609. English, Portuguese. PMID 32901659
- [Background] Plunkett A, McCoart A, Howard RS, Dennison E, Bartoszek M. A randomized, single-blind, prospective trial of auricular 'battlefield' acupuncture for the reduction of postoperative tonsillectomy pain in adults. Pain Manag. 2018 Jul 1;8(4):287-295. doi: 10.2217/pmt-2018-0007. Epub 2018 Jun 14. PMID 29898645
- [Background] Wan LS, Li WS, Li WY, Li GC. [Observation on the anesthesia effect of general anesthesia assisted by auricular-plaster therapy in gynecological surgery]. Zhongguo Zhen Jiu. 2013 Mar;33(3):237-40. Chinese. PMID 23713310
- [Background] Michalek-Sauberer A, Heinzl H, Sator-Katzenschlager SM, Monov G, Knolle E, Kress HG. Perioperative auricular electroacupuncture has no effect on pain and analgesic consumption after third molar tooth extraction. Anesth Analg. 2007 Mar;104(3):542-7. doi: 10.1213/01.ane.0000253233.51490.dd. PMID 17312205
- [Background] Alimi D, Chelly JE. New Universal Nomenclature in Auriculotherapy. J Altern Complement Med. 2018 Jan;24(1):7-14. doi: 10.1089/acm.2016.0351. Epub 2017 Aug 23. PMID 28832182
- [Background] Alimi D, Geisdsmann A, Gardeur D. Auricular acupuncture stimulation measured on functional magnetic Imaging. Med Acup 2002;13:18-21
- [Background] Romoli M, Allais G, Airola G, Benedetto C, Mana O, Giacobbe M, Pugliese AM, Battistella G, Fornari E. Ear acupuncture and fMRI: a pilot study for assessing the specificity of auricular points. Neurol Sci. 2014 May;35 Suppl 1:189-93. doi: 10.1007/s10072-014-1768-7. PMID 24867864
- [Background] Alimi, D. L'Auriculotherapie Medicale: Bases Scientifiques. Principles, Indications et Strategies Therapeutiques. Elsevier Masson SAS, 2017. pp 87-99. French
- [Background] Wirz-Ridolfi A. The History of Ear Acupuncture and Ear Cartography: Why Precise Mapping of Auricular Points Is Important. Med Acupunct. 2019 Jun 1;31(3):145-156. doi: 10.1089/acu.2019.1349. Epub 2019 Jun 17. PMID 31297168
- [Background] Alimi, D. L'Auriculotherapie Medicale: Bases Scientifiques, Principles, Indications et Strategies Therapeutiques. Chapitre 10. Neurophysiologie des perceptions. Elsevier Masson
- [Background] Felten DL, Shetty AN. Second edition of the Netter's Atlas of Neuroscience Chapter 9. Peripheral nervous system. Publisher Saunders, Elsevier;2010. pp 135-172
- [Background] Peuker ET, Filler TJ. The nerve supply of the human auricle. Clin Anat. 2002 Jan;15(1):35-7. doi: 10.1002/ca.1089. PMID 11835542
- [Background] Anthwal N, Thompson H. The development of the mammalian outer and middle ear. J Anat. 2016 Feb;228(2):217-32. doi: 10.1111/joa.12344. Epub 2015 Jul 30. PMID 26227955
- [Background] Rouwette T, Vanelderen P, Roubos EW, Kozicz T, Vissers K. The amygdala, a relay station for switching on and off pain. Eur J Pain. 2012 Jul;16(6):782-92. doi: 10.1002/j.1532-2149.2011.00071.x. Epub 2011 Dec 19. PMID 22337528
- [Background] Babygirija R, Sood M, Kannampalli P, Sengupta JN, Miranda A. Percutaneous electrical nerve field stimulation modulates central pain pathways and attenuates post-inflammatory visceral and somatic hyperalgesia in rats. Neuroscience. 2017 Jul 25;356:11-21. doi: 10.1016/j.neuroscience.2017.05.012. Epub 2017 May 17. PMID 28526575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the pre-operative holding area of UPMC Shadyside or UPMC Montefiore Hospitals on the day of their scheduled rotator cuff surgery. Recruitment began on January 24, 2020 and concluded on July 1, 2021. During this time, recruitment was on hold due to COVID-19 protocol from February to July of 2020.
Pre-assignment Details: A total of 50 subjects signed an informed consent and all subjects were randomized to either the placebo or intervention group. No subjects were excluded prior to randomization.
Period: Overall Study
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Started | 25 | 25
Completed | 19 | 20
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 5 | 5
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Groups:
- Total: Total of all reporting groups
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.5) | 61.4 (9.9) | 61.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Height [Mean (Standard Deviation); unit: centimeters] | 170.2 (12.4) | 169.1 (10.2) | 169.6 (11.0)
Weight [Mean (Standard Deviation); unit: kilograms] | 85.9 (17.8) | 94.7 (27.2) | 90.3 (23.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (3.6) | 32.8 (7.5) | 31.2 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption Following Rotator Cuff Surgery
Description: Investigate the efficacy of auriculotherapy in reducing perioperative opioid consumption in opioid-naïve patients undergoing elective rotator cuff surgery. This is reported in consumption of oral morphine mg equivalents (OME) at 24 hrs, 48 hrs, 72 hrs, 96 hrs, and 120 hrs post-operative as well as the total sum of these intervals
Time Frame: 24 hrs, 48 hrs, 72 hrs, 96 hrs, and 120 hrs post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: oral morphine mg equivalents (OME)
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
oral morphine mg equivalents (OME)
  24 Hours | 31 (20) | 25 (20)
  48 Hours | 25 (17) | 21 (17)
  72 Hours | 19 (19) | 12 (13)
  96 Hours | 12 (15) | 9 (10)
  120 Hours | 10 (13) | 5 (7)
  Total | 96 (67) | 62 (46)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 24 hrs; Test type: Superiority; p = 0.1771, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 2: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 48 hrs; Test type: Superiority; p = 0.2833, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 3: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 72 hrs; Test type: Superiority; p = 0.0909, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 4: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 96 hrs; Test type: Superiority; p = 0.2310, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 5: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 120 hrs; Test type: Superiority; p = 0.0801, t-test, 1 sided
Statistical Analysis 6: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Total; Test type: Superiority; p = 0.0307, t-test, 1 sided — P value less than 0.1 will be considered significant

2. Secondary Outcome: Post-Operative Pain With Movement
Description: Numerical Rating Scale (NRS) Pain with movement on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a worse outcome.
Time Frame: 24 hrs through 90-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
score on a scale
  24 Hours | 8.11 (2.11) | 7.42 (2.67)
  48 Hours | 6.83 (2.28) | 6.21 (2.70)
  72 Hours | 6.28 (2.19) | 5.37 (2.22)
  96 Hours | 5.44 (2.59) | 4.65 (2.30)
  120 Hours | 4.72 (2.61) | 3.80 (2.28)
  Day 14 | 5.84 (2.39) | 4.47 (2.12)
  Day 30 | 5.00 (2.78) | 5.27 (2.84)
  Day 60 | 4.15 (3.48) | 3.64 (2.90)
  Day 90 | 2.21 (1.85) | 2.00 (2.61)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 24 hrs; Test type: Superiority; p = 0.1956, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 2: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 48 hrs; Test type: Superiority; p = 0.2274, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 3: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 72 hrs; Test type: Superiority; p = 0.1090, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 4: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 96 hrs; Test type: Superiority; p = 0.1618, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 5: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 120 hrs; Test type: Superiority; p = 0.1264, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 6: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 14; Test type: Superiority; p = 0.0394, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 7: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 30; Test type: Superiority; p = 0.3968, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 8: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 60; Test type: Superiority; p = 0.3407, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 9: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 90; Test type: Superiority; p = 0.4033, t-test, 1 sided — P value less than 0.1 will be considered significant

3. Secondary Outcome: Post-Operative Pain at Rest
Description: Numerical Rating Scale (NRS) pain at rest on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a worse outcome.
Time Frame: Time of discharge through 90-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
score on a scale
  Discharge | 0.89 (1.91) | 0.45 (0.76)
  24 Hours | 6.17 (3.01) | 5.75 (3.32)
  48 Hours | 4.67 (3.18) | 4.50 (2.69)
  72 Hours | 3.89 (2.72) | 3.50 (2.19)
  96 Hours | 3.50 (2.41) | 3.45 (2.44)
  120 Hours | 2.88 (2.00) | 2.65 (2.28)
  Day 14 | 2.26 (1.59) | 1.71 (1.76)
  Day 30 | 2.13 (2.00) | 1.20 (1.37)
  Day 60 | 1.23 (2.05) | 1.21 (1.67)
  Day 90 | 0.43 (0.76) | 0.38 (0.77)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Time of discharge; Test type: Superiority; p = 0.1707, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 2: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 24 hrs; Test type: Superiority; p = 0.3446, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 3: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 48 hrs; Test type: Superiority; p = 0.4310, t-test, 1 sided
Statistical Analysis 4: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 72 hrs; Test type: Superiority; p = 0.3143, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 5: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 96 hrs; Test type: Superiority; p = 0.4749, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 6: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 120 hrs; Test type: Superiority; p = 0.3728, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 7: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 14; Test type: Superiority; p = 0.1628, t-test, 1 sided
Statistical Analysis 8: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 30; Test type: Superiority; p = 0.0731, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 9: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 60; Test type: Superiority; p = 0.4909, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 10: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 90; Test type: Superiority; p = 0.4411, t-test, 1 sided — P value less than 0.1 will be considered significant

4. Secondary Outcome: Non-narcotic Analgesic Consumption
Description: Investigate the efficacy of auriculotherapy in reducing total perioperative consumption of non-narcotic analgesics.
Time Frame: Day of surgery through 5-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
milligrams
  Acetaminophen | 4438.16 (4066.01) | 5955.63 (5882.27)
  Ibuprofen | 785.26 (1576.68) | 1370.00 (2386.17)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Acetaminophen; Test type: Superiority; p = 0.1786, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 2: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Ibuprofen; Test type: Superiority; p = 0.1876, t-test, 1 sided — P value less than 0.1 will be considered significant

5. Secondary Outcome: Functional Recovery Questionnaire 12-Item Short Form Health Survey (SF-12)
Description: Functional recovery will be measured by the assessment of the participant's answers to the Functional Recovery Questionnaire 12-Item Short Form Health Survey (SF-12). The SF-12 Health Survey includes questions from the SF-36 Health Survey (Version 1). Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average. The highest possible PCS-12 score is 56.57706 and the lowest possible score is 23.99938. The highest possible MCS-12 score is 67.37178 and the lowest possible score is 17.57825. Higher scores for both represent better functioning.
Time Frame: Day of surgery through 90 days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
score on a scale
  Baseline PCS | 38.9 (8.4) | 38.0 (6.6)
  Day 14 PCS | 37.1 (8.2) | 34.0 (4.6)
  Day 30 PCS | 36.1 (7.6) | 35.7 (4.7)
  Day 60 PCS | 40.5 (9.2) | 39.0 (8.4)
  Day 90 PCS | 44.1 (8.4) | 44.9 (7.8)
  Baseline MCS | 60.5 (4.4) | 59.4 (3.8)
  Day 14 MCS | 57.4 (8.1) | 60.3 (5.3)
  Day 30 MCS | 61.3 (5.1) | 59.6 (4.6)
  Day 60 MCS | 59.9 (5.5) | 58.6 (3.9)
  Day 90 MCS | 60.8 (2.5) | 58.3 (4.7)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Baseline PCS; Test type: Superiority; p = 0.3638, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 2: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 14 PCS; Test type: Superiority; p = 0.0856, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 3: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 30 PCS; Test type: Superiority; p = 0.4428, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 4: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 60 PCS; Test type: Superiority; p = 0.3378, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 5: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 90 PCS; Test type: Superiority; p = 0.3942, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 6: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Baseline MCS; Test type: Superiority; p = 0.2190, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 7: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 14 MCS; Test type: Superiority; p = 0.1112, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 8: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 30 MCS; Test type: Superiority; p = 0.1737, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 9: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 60 MCS; Test type: Superiority; p = 0.2408, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 10: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 90 MCS; Test type: Superiority; p = 0.0380, t-test, 1 sided — P value less than 0.1 will be considered significant

6. Secondary Outcome: Length of Recovery Room Stay
Description: Evaluate time to readiness for discharge from post-anesthesia care unit (PACU) from out of OR time in minutes
Time Frame: Day of surgery through recovery room discharge, up to 142 min post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
minutes | 59.5 (25.7) | 67.2 (34.1)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Test type: Superiority; p = 0.2220, t-test, 1 sided — P value less than 0.1 will be considered significant

7. Secondary Outcome: Length of Hospital Stay
Description: Evaluate time to hospital discharge from out of OR time in minutes
Time Frame: Day of surgery through time of discharge, up to 270 min post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
minutes | 140.1 (32.1) | 148.0 (47.4)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Test type: Superiority; p = 0.2856, t-test, 1 sided — P value less than 0.1 will be considered significant

8. Secondary Outcome: Number of Participants Who Experienced Post-operative Complications
Description: The number of participants who experienced complications and received the standard protocol versus subjects who received the standard protocol + Auriculotherapy. Post-operative complications can be defined as unexpected problems that arise following surgery including increased bleeding, infection, recurrent rotator cuff tear, and displacement of suture anchor.
Time Frame: Day of surgery through 90-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

9. Secondary Outcome: Subjects Requiring Readmission Due to Pain
Description: Evaluate the number of subjects readmitted because of pain or pain-related issues during the 90 day study duration
Time Frame: Day of surgery through 90-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Number; unit: participants
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
participants | 0 | 0

10. Secondary Outcome: Overall Patient Satisfaction
Description: Participants are asked to assess their overall satisfaction with care upon discharge on a 10-point satisfaction scale of 0 (least satisfaction) to 10 (highest satisfaction). The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a better outcome.
Time Frame: Day of surgery through time of discharge, up to 270 min post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
score on a scale | 9.2 (2.1) | 9.6 (0.6)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Test type: Superiority; p = 0.2241, t-test, 1 sided

11. Secondary Outcome: Satisfaction With Pain Management
Description: Participants are asked to assess their satisfaction with pain management at discharge, 24 hrs, 48 hrs, 72 hrs, 96, hours, 120 hrs and 14 days, 30 days, 60 days and 90 days post-operative on a 10-point satisfaction scale of 0 (least satisfaction) to 10 (highest satisfaction). The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a better outcome.
Time Frame: Day of surgery through 90-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
score on a scale
  Discharge | 5.7 (0.7) | 5.9 (0.4)
  24 Hours | 4.2 (1.8) | 4.1 (1.4)
  48 Hours | 4.7 (1.2) | 4.6 (1.1)
  72 Hours | 5.1 (0.8) | 4.9 (1.0)
  96 Hours | 4.7 (1.5) | 4.6 (1.3)
  120 Hours | 4.8 (1.5) | 4.8 (1.1)
  Day 14 | 5.6 (0.8) | 5.6 (0.8)
  Day 30 | 5.4 (1.2) | 5.7 (0.5)
  Day 60 | 5.2 (1.6) | 5.3 (1.5)
  Day 90 | 4.9 (1.9) | 5.9 (0.3)
Statistical Analysis 1: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Time of discharge; Test type: Superiority; p = 0.2714, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 2: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 24 hrs; Test type: Superiority; p = 0.3749, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 3: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 48 hrs; Test type: Superiority; p = 0.3862, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 4: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 72 hrs; Test type: Superiority; p = 0.1735, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 5: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 96 hrs; Test type: Superiority; p = 0.4304, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 6: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; 120 hrs; Test type: Superiority; p = 0.4902, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 7: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 14; Test type: Superiority; p = 0.4371, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 8: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 30; Test type: Superiority; p = 0.1950, t-test, 1 sided — P value less than 0.1 will be considered significant
Statistical Analysis 9: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 60; Test type: Superiority; p = 0.4124, t-test, 1 sided
Statistical Analysis 10: Comparison: Auriculotherapy Without Nitrogen Gas vs Auriculotherapy With Nitrogen Gas; Day 90; Test type: Superiority; p = 0.0268, t-test, 1 sided — P value less than 0.1 will be considered significant

12. Secondary Outcome: Subjects Requiring Hospital Readmission
Description: Evaluate the number of subjects readmitted to the hospital for post-operative complications other than pain-related issues.
Time Frame: Day of surgery through 90-days post-operative
Population: Patients undergoing elective rotator cuff repair with an interscalene block and general anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the subject's participation in the study (90 days post-operative).
Description: Adverse event data was collected for the duration of the subject's 90-day study participation using the electronic medical record and via patient report at day 5, 14, 30, 60, and 90 follow-ups.
Arm/Group | Auriculotherapy Without Nitrogen Gas | Auriculotherapy With Nitrogen Gas
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/19 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auriculotherapy Without Nitrogen Gas (N=19) | Auriculotherapy With Nitrogen Gas (N=20)
Postoperative Constipation (Gastrointestinal disorders) | 4 (4) | 10 (10) — Constipation is infrequent bowel movements or difficult passage of stools that persists for several days to weeks

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03860259/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03860259/ICF_001.pdf